CLINICAL TRIAL: NCT04677985
Title: Menthol-based Topical Analgesic Induces Similar Upper and Lower Body Increases in Pain Pressure Threshold: A Randomized Trial
Brief Title: Analgesic Induces Similar Upper and Lower Body Pain Pressure Threshold Increases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, David George Behm, University Research Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20192544
Record Dates: First submitted 2020-12-14; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Pain, Acute; Muscle Soreness; Tendon Injuries
Keywords: menthol; musculoskeletal; tendons; lower back
MeSH Terms: conditions — Acute Pain; Myalgia; Tendon Injuries

STUDY DESIGN:
Intervention Model Description: Random allocation of the application of a menthol based topical analgesic versus a placebo.
Who Masked: Participant, Investigator
Masking Description: Placebo and analgesic applications were identified by numbers which were only revealed after the statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol based topical analgesic (Experimental): Menthol based topical analgesic was applied to a variety of upper and lower body muscles and tendons.
  Interventions: Combination Product: Menthol based topical analgesic
- Placebo (Placebo Comparator): Placebo (cream that smelled like menthol) was applied to a variety of upper and lower body muscles and tendons.
  Interventions: Combination Product: Menthol based topical analgesic

INTERVENTIONS:
Combination Product: Menthol based topical analgesic — Topical analgesic or placebo was applied to upper and lower body muscles and tendons and pain pressure threshold was measured with a handheld algometer.
  Other Names: Menthol smelling cream with no analgesic

SUMMARY:
Background: Both health professionals and consumers use menthol-based topical analgesics extensively for the temporary relief of pain from musculoskeletal ailments or injury. However, there are no reports of differences in the pain pressure threshold (PPT) or the relative effectiveness of topical analgesics to reduce pain in the upper and lower body muscles and tendons. Objectives: The objective of this study was to investigate whether differences existed in PPT and relative pain attenuation associated with a menthol based topical analgesic over a variety of upper and lower body muscles and tendons. Design: Randomized allocation, controlled, intervention study. Method: Sixteen participants (10 females and 6 males), who were tested on their dominant or non-dominant side. The order of specific muscle / tendon testing was also randomized, which included upper body (middle deltoid, biceps brachii, and lateral epicondylar tendon) and lower body locations (quadriceps, hamstrings, gastrocnemius, lumbo-sacral erector spinae muscles, and patellar and Achilles tendons). PPT was monitored before and 15-minutes following the application of a menthol based topical analgesic.

DETAILED DESCRIPTION:
Experimental Design Using random allocation (slip of paper chosen from a box by one of the researchers), participants were either tested on their dominant or non-dominant side. Limb dominance was determined by the participants' self-report of the preferred hand used for writing/throwing (upper extremity) and for kicking a ball (lower extremity). Further, randomization was used to determine which muscle groups would be tested first: upper body versus lower body, and the order of muscle testing. The tested upper body limb muscles consisted of the middle deltoid, and biceps brachii. The lower body muscle groups consisted of the quadriceps, hamstrings, and gastrocnemius. In order to compare sensitivity differences between muscles and tendons, the patellar tendon, and Achilles tendon were also tested. In addition, as tennis elbow (lateral epicondylitis/epicondylosis) is a common injury [40], the lateral epicondylar tendon was also evaluated. The lower back was tested using the lumbo-sacral erector spinae muscles.

The pre-testing consisted of obtaining PPT (without topical analgesic application) using a handheld algometer (Lafayette Manual Muscle Test System™, Model 01163, Lafayette Instrument Company, Indiana, USA), from each muscle or tendon. The algometer was a hand-held muscle tester with a range of 0-300 pounds (136.1 kilograms) that consisted of a padded disc with a surface area of 1.7 cm2 attached to a microprocessor-control unit that measures peak force (pounds or kilograms). The unit has a digital readout for peak-applied pressure and provides a built-in calibration routine that verifies a valid calibration. The pain threshold was defined as the minimum pressure that induced pain [15]. Participants were instructed to provide a verbal report as soon as the quality of sensation changed from pressure to pain [15,16] at which point the algometer was removed. This study chose to measure the PPT via a pressure algometer as it has been shown to be a clinically and experimentally reliable method to assess pain [16,23,35]. The middle of the muscle belly for the biceps brachii, middle deltoid, hamstrings (biceps femoris), quadriceps (rectus femoris), and gastrocnemius was used. The measurement sites for the patella tendon and lateral epicondylar tendon were 1 cm distal from the bony origin. For the Achilles tendon, the measurement was taken at one third of the distance of the tendon length distal to its insertion. There were three readings from each testing position with a 5-second rest period between each reading.

Intervention The intervention involved the application of 4% menthol-based Biofreeze® (Performance Health, Akron, Ohio) to the muscles and tendons immediately following the pre-testing. Based on prior recommendations [22,45,32] varying volumes of the topical analgesic were applied in reference to the surface area of the muscle. The previously cited investigators recommended 1ml per 200 cm2 of muscle surface area. No significant force (light stroking actions to apply the analgesic) was used for the application of the menthol-based topical analgesic.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals with no musculoskeletal or neural pathologies.

Exclusion Criteria:

1. Musculoskeletal or neural pathologies / injuries in the year before the experiment.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | Applied 15 minutes after application of topical analgesic or placebo.
  Measures the force applied to the muscle or tendon till pain is detected.

CONTACTS AND LOCATIONS:
Overall Officials: David G Behm, PhD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: Yes
Excel sheet data can be obtained upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 14, 2020 onwards